CLINICAL TRIAL: NCT04434131
Title: Open, Non-comparative Pilot Study to Provide Access to Treatment With Investigational Convalescent Plasma and Measure Antibody Levels in Patients Hospitalized With COVID-19
Brief Title: Treatment With Investigational Convalescent Plasma and Measure Antibody Levels in Patients Hospitalized With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Michelle Harkins, Division Chief of Pulmonary/ Critical Care/Sleep Medicine, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-227
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Results first posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Convalescent Plasma (Experimental): The investigational product is anti-SARS-CoV-2 convalescent plasma obtained from former patients identified as having recovered from COVID-19 and obtained by Vitalant from local and national donors following national blood donation guidelines. All subjects receive the convalescent plasma.
  Interventions: Drug: Convalescent Plasma

INTERVENTIONS:
Drug: Convalescent Plasma — Study subjects will receive 1 unit (200mL) of SARS-CoV-2 convalescent plasma collected from a single donor who recovered from COVID-19.
  Other Names: Not appicable

SUMMARY:
This is an open label pilot study designed to provide access to treatment with investigational convalescent plasma and assess the relationship between NAb titers in the investigational convalescent plasma compared to changes in NAb levels in the recipient in hospitalized patients with COVID-19.

DETAILED DESCRIPTION:
Primary objectives are as follows:

1. To provide access to treatment with investigational convalescent plasma to inpatients with documented COIVD-19 infection
2. To measure NAb titers in an aliquot of the CP administered, to measure the volume of CP administered, and determine whether there is a correlation between the NAb dose (in NAb units/kg body weight, where a unit is the reciprocal of the endpoint NAb titer in the CP multiplied by the volume in ml) and change or lack of change when comparing pre-treatment and day one NAb titers.

Secondary, exploratory objectives are as follows:

1. To evaluate the safety of convalescent plasma (CP) administration in hospitalized COVID-19 patients
2. To evaluate viral shedding of SARSCoV-2 in nasopharyngeal or nasal samples before and on days 3, 7, and 14 after CP transfusion
3. To perform genomic analysis of the SARS-CoV-2 from patients before and after treatment with CP transfusion
4. Determine cumulative incidence of disease severity (transfer to ICU, type of respiratory support, LOS, and mortality)

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older.
2. Hospitalized with COVID-19 respiratory symptoms and confirmation via COVID-19 SARS-CoV-2 RT-PCR testing. If COVID-19 test results are pending or done at enrolment, test results must be positive prior to administration of convalescent plasma.
3. Patient (or legally authorized representative, LAR) is willing and able to provide written informed consent and comply with all protocol requirements.
4. For patients unable to consent, consent by the legally authorized representative (LAR) may be obtained by phone.

Exclusion Criteria:

1. Female subjects with positive pregnancy test or breastfeeding.
2. Receipt of pooled immunoglobulin in past 30 days.
3. Contraindication to transfusion or history of prior severe allergic reactions to transfused blood products.
4. On ECMO or in refractory shock at entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969
- [Derived] Chai KL, Valk SJ, Piechotta V, Kimber C, Monsef I, Doree C, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2020 Oct 12;10:CD013600. doi: 10.1002/14651858.CD013600.pub3. PMID 33044747
- [Derived] Bradfute SB, Hurwitz I, Yingling AV, Ye C, Cheng Q, Noonan TP, Raval JS, Sosa NR, Mertz GJ, Perkins DJ, Harkins MS. Severe Acute Respiratory Syndrome Coronavirus 2 Neutralizing Antibody Titers in Convalescent Plasma and Recipients in New Mexico: An Open Treatment Study in Patients With Coronavirus Disease 2019. J Infect Dis. 2020 Oct 13;222(10):1620-1628. doi: 10.1093/infdis/jiaa505. PMID 32779705

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: The investigational product is anti-SARS-CoV-2 convalescent plasma obtained from former patients identified as having recovered from COVID-19 and obtained by Vitalant from local and national donors following national blood donation guidelines. All subjects receive the convalescent plasma.
  Convalescent Plasma: Study subjects will receive 1 unit (200mL) of SARS-CoV-2 convalescent plasma collected from a single donor who recovered from COVID-19.
Period: Overall Study
Arm/Group | Single Arm
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 52 [39 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: NAb Dose Titer in the Convalescent Plasma (CP), Pre-treatment, and Day One in Hospitalized Patients With Documented COVID-19 Infection
Description: Neutralizing antibody titer (PRNT 80)
Time Frame: Day of convalescent plasma infusion (day 0) and following day (day 1)
Population: Participants were hospitalized patients receiving CP and donors were not considered participants of the study. Again, 12 donors contributed to CP but were not enrolled in the study. Mean titer from donor CP obtained from 12 donors.
Measure: Mean (Standard Error); unit: titer
Arm/Group | Single Arm
Number analyzed (Participants) | 12
titer
  Donor convalescent plasma | 56.7 (32.4)
  Day 0 (pre-treatment in hospitalized patients) | 390 (369)
  Day 1 (in hospitalized patients) | 413 (363)

2. Secondary Outcome: Number of Participants With Rapid Deterioration as Evidenced by Increase in Ordinal Score
Description: World Health Organization ordinal scale, with scores defined as follows: 5, hospitalized, requiring any supplemental oxygen; 6, hospitalized, requiring noninvasive ventilation or use of high-flow oxygen devices; 7, hospitalized, receiving invasive mechanical ventilation or extracorporeal membrane oxygenation; and 8, death.
Time Frame: Within 4 hours of transfusion
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 12
Participants | 0

3. Secondary Outcome: Number of Participants With Clearance of Viral Shedding of SARS CoV-2 in Nasopharyngeal Samples
Time Frame: Day 0,1,3,7 and 14
Population: Data was not collected
Arm/Group | Single Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/31/NCT04434131/Prot_SAP_001.pdf
  • Informed Consent Form (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT04434131/ICF_000.pdf